CLINICAL TRIAL: NCT02697591
Title: A Phase 1/2, Open-Label, Dose-Escalation, Safety and Tolerability Study of INCAGN01876 in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: A Study of INCAGN01876 in Participants With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Biosciences International Sàrl (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCAGN 1876-101
Record Dates: First submitted 2016-02-22; First posted 2016-03-03 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Advanced Malignancies; Metastatic Cancer
Keywords: Solid tumor; adenocarcinoma of the endometrium; melanoma, non-small cell lung cancer (NSCLC); renal cell carcinoma (RCC); glucocorticoid-induced tumor necrosis factor receptor (GITR)
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Phase 1: 20.0 Milligram Per Kilograms (mg/kg) Every 2 Weeks (Q2W) (Experimental): Participants received IV infusion of study drug at a dose of 20.0 mg/kg every Q2W starting on Day 1 of each cycle for up to 15 months.
  Interventions: Drug: INCAGN01876
- Phase 1: 0.03 mg/kg Q2W (Experimental): Participants received intravenous (IV) infusion of study drug at a dose of 0.03 mg/kg every Q2W starting on Day 1 of each cycle for up to 15 months.
  Interventions: Drug: INCAGN01876
- Phase 1: 0.1 mg/kg Q2W (Experimental): Participants received IV infusion of study drug at a dose of 0.1 mg/kg every Q2W starting on Day 1 of each cycle for up to 15 months.
  Interventions: Drug: INCAGN01876
- Phase 1: 0.3 mg/kg Q2W (Experimental): Participants received IV infusion of study drug at a dose of 0.3 mg/kg every Q2W starting on Day 1 of each cycle for up to 15 months.
  Interventions: Drug: INCAGN01876
- Phase 1: 1.0 mg/kg Q2W (Experimental): Participants received IV infusion of study drug at a dose of 1.0 mg/kg every Q2W starting on Day 1 of each cycle for up to 15 months.
  Interventions: Drug: INCAGN01876
- Phase 1: 3.0 mg/kg Q2W (Experimental): Participants received IV infusion of study drug at a dose of 3.0 mg/kg every Q2W starting on Day 1 of each cycle for up to 15 months.
  Interventions: Drug: INCAGN01876
- Phase 1: 5.0 mg/kg Q2W (Experimental): Participants received IV infusion of study drug at a dose of 5.0 mg/kg every Q2W starting on Day 1 of each cycle for up to 15 months.
  Interventions: Drug: INCAGN01876
- Phase 1: 10.0 mg/kg Q2W (Experimental): Participants received IV infusion of study drug at a dose of 10.0 mg/kg every Q2W starting on Day 1 of each cycle for up to 15 months.
  Interventions: Drug: INCAGN01876
- Phase 1: 400 mg/kg Every 4 Weeks (Q4W) (Experimental): Participants received IV infusion of study drug at a dose of 400 mg/kg every Q2W starting on Day 1 of each cycle for up to 15 months.
  Interventions: Drug: INCAGN01876
- Phase 2: 300 mg/kg Q2W (Experimental): Participants received IV infusion of study drug at a dose of 300 mg/kg every Q2W starting on Day 1 of each cycle for up to 15 months.
  Interventions: Drug: INCAGN01876

INTERVENTIONS:
Drug: INCAGN01876 — Initial cohort dose of INCAGN01876 monotherapy at the protocol-defined starting dose, with subsequent cohort escalations based on protocol-specific criteria. The recommended dose will be taken forward into expansion cohorts.

SUMMARY:
This was an open-label, non-randomized Phase 1/2 safety study of INCAGN01876 in participants with advanced or metastatic solid tumors that was conducted in 2 parts. Part 1 is dose escalation and safety expansion which determines the optimal dose and maximum number of tolerated doses. Part 2 is dose expansion in which Part 1 recommended dose will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic disease; locally advanced disease must not be amenable to resection with curative intent.
* Part 1: Participants with advanced or metastatic solid tumors.
* Part 2: Participants with advanced or metastatic adenocarcinoma of endometrium, melanoma, non-small cell lung cancer, and renal cell carcinoma.
* Participants who have disease progression after treatment with available therapies that are known to confer clinical benefit, or who are intolerant to treatment, or participants who refuse standard treatment.
* Presence of measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.

Exclusion Criteria:

* Laboratory and medical history parameters not within the protocol-defined range.
* Receipt of anticancer medications or investigational drugs within protocol-defined intervals before the first administration of study drug.
* Has not recovered to ≤ Grade 1 from toxic effects of prior therapy and/or complications from prior surgical intervention before starting therapy.
* Receipt of a live vaccine within 30 days of planned start of study therapy.
* Active autoimmune disease.
* Prior treatment with any tumor necrosis factor super family agonist.
* Known active central nervous system metastases and/or carcinomatous meningitis.
* Evidence of active, non-infectious pneumonitis or history of interstitial lung disease.
* Evidence of hepatitis B virus or hepatitis C virus infection or risk of reactivation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Janik, MD, Study Director — Incyte Corporation
Locations (8):
- United States (8):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering at Monmouth, Middletown, New Jersey
  - MSK Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamid O, Cardin DB, Hodi FS, LoRusso P, Merghoub T, Zappasodi R, Maniyar R, Janik JE, van der Velden MVW, Zhou F, Dong Z, Chen X, Harding JJ. First-in-Human Phase I/II Study of INCAGN01876, a Glucocorticoid-Induced Tumor Necrosis Factor Receptor Agonist, in Patients with Advanced or Metastatic Solid Tumors. Clin Cancer Res. 2025 Oct 1;31(19):4089-4100. doi: 10.1158/1078-0432.CCR-24-4141. PMID 40711469

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 100 participants were enrolled at 7 study sites in the United States from 20 June 2016 to 16 December 2019.
Groups:
- Phase 1: 0.03 mg/kg Q2W: Participants received intravenous (IV) infusion of study drug at a dose of 0.03 mg/kg Q2W starting on Day 1 of each cycle for up to 15 months.
- Phase 1: 0.1 mg/kg Q2W: Participants received IV infusion of study drug at a dose of 0.1 mg/kg Q2W starting on Day 1 of each cycle for up to 15 months.
- Phase 1: 0.3 mg/kg Q2W: Participants received IV infusion of study drug at a dose of 0.3 mg/kg Q2W starting on Day 1 of each cycle for up to 15 months.
- Phase 1: 1.0 mg/kg Q2W: Participants received IV infusion of study drug at a dose of 1.0 mg/kg Q2W starting on Day 1 of each cycle for up to 15 months.
- Phase 1: 3.0 mg/kg Q2W: Participants received IV infusion of study drug at a dose of 3.0 mg/kg Q2W starting on Day 1 of each cycle for up to 15 months.
- Phase 1: 5.0 mg/kg Q2W: Participants received IV infusion of study drug at a dose of 5.0 mg/kg Q2W starting on Day 1 of each cycle for up to 15 months.
- Phase 1: 10.0 mg/kg Q2W: Participants received IV infusion of study drug at a dose of 10.0 mg/kg Q2W starting on Day 1 of each cycle for up to 15 months.
- Phase 1: 20.0 mg/kg Q2W: Participants received IV infusion of study drug at a dose of 20.0 mg/kg Q2W starting on Day 1 of each cycle for up to 15 months.
- Phase 1: 400 mg Q4W: Participants received IV infusion of study drug at a dose of 400 mg Q4W starting on Day 1 of each cycle for up to 15 months.
- Phase 2: 300 mg Q2W: Participants received IV infusion of study drug at a dose of 300 mg Q2W starting on Day 1 of each cycle for up to 15 months.
Period: Overall Study
Arm/Group | Phase 1: 0.03 mg/kg Q2W | Phase 1: 0.1 mg/kg Q2W | Phase 1: 0.3 mg/kg Q2W | Phase 1: 1.0 mg/kg Q2W | Phase 1: 3.0 mg/kg Q2W | Phase 1: 5.0 mg/kg Q2W | Phase 1: 10.0 mg/kg Q2W | Phase 1: 20.0 mg/kg Q2W | Phase 1: 400 mg Q4W | Phase 2: 300 mg Q2W
Started | 4 | 4 | 4 | 3 | 15 | 18 | 16 | 4 | 10 | 22
Completed | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 2
Not Completed | 4 | 4 | 3 | 3 | 13 | 16 | 16 | 3 | 9 | 20
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 1 | 7 | 6 | 9 | 1 | 6 | 10
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1
Not completed — Death | 2 | 3 | 1 | 1 | 4 | 5 | 3 | 1 | 1 | 5
Not completed — Reason not Specified | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants enrolled in the study who received at least 1 dose of study drug.
Groups:
- Phase 1: 0.03 mg/kg Q2W: INCAGN01876 was administered at 0.03mg/kg Q2W as part of dose escalation.
- Phase 1: 0.1 mg/kg Q2W: INCAGN01876 was administered at 0.1mg/kg Q2W as part of dose escalation.
- Phase 1: 0.3 mg/kg Q2W: INCAGN01876 was administered at 0.3mg/kg Q2W as part of dose escalation.
- Phase 1: 1.0 mg/kg Q2W: INCAGN01876 was administered at 1.0mg/kg Q2W as part of dose escalation.
- Phase 1: 3.0 mg/kg Q2W: INCAGN01876 was administered at 3mg/kg Q2W as part of dose escalation.
- Phase 1: 5.0 mg/kg Q2W: INCAGN01876 was administered at 5mg/kg Q2W as part of dose escalation.
- Phase 1: 10.0 mg/kg Q2W: INCAGN01876 was administered at 10mg/kg Q2W as part of dose escalation.
- Phase 1: 20.0 mg/kg Q2W: INCAGN01876 was administered at 20mg/kg Q2W as part of dose escalation.
- Phase 1: 400 mg Q4W: INCAGN01876 was administered at 400mg Q4W as part of dose escalation.
- Phase 2: 300 mg Q2W: INCAGN01876 was administered at 300mg Q2W as part of dose escalation.
- Total: Total of all reporting groups
Arm/Group | Phase 1: 0.03 mg/kg Q2W | Phase 1: 0.1 mg/kg Q2W | Phase 1: 0.3 mg/kg Q2W | Phase 1: 1.0 mg/kg Q2W | Phase 1: 3.0 mg/kg Q2W | Phase 1: 5.0 mg/kg Q2W | Phase 1: 10.0 mg/kg Q2W | Phase 1: 20.0 mg/kg Q2W | Phase 1: 400 mg Q4W | Phase 2: 300 mg Q2W | Total
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 15 | 18 | 16 | 4 | 10 | 22 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (17.02) | 45.3 (21.01) | 70.0 (12.19) | 53.0 (14.93) | 62.3 (10.58) | 53.6 (12.83) | 62.3 (10.22) | 59.5 (14.75) | 57.6 (12.02) | 67.2 (10.86) | 60.1 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 0 | 8 | 7 | 5 | 1 | 4 | 10 | 42
  Male | 2 | 1 | 2 | 3 | 7 | 11 | 11 | 3 | 6 | 12 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 5
  Ethnicity: Not Hispanic or Latino | 4 | 4 | 4 | 3 | 14 | 16 | 15 | 4 | 9 | 19 | 92
  Ethnicity: Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Ethnicity: Unknown | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Caucasian | 3 | 3 | 2 | 2 | 13 | 15 | 12 | 4 | 7 | 21 | 82
  Race: Black/African-American | 1 | 1 | 1 | 0 | 2 | 1 | 2 | 0 | 0 | 1 | 9
  Race: Asian | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 5
  Race: Missing | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 4
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used to assess how a participant's disease is progressing and assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. Graded from 0-5 where 0=Fully Active (Most Favorable Activity); 1=Restricted activity but ambulatory; 2=Ambulatory but unable to carry out work activities; 3=Limited Self-Care; 4=Completely Disabled, No self-care; 5=Dead (Least Favorable Activity).
  Participants
    0 | 3 | 1 | 3 | 2 | 8 | 10 | 8 | 1 | 6 | 12 | 54
    1 | 1 | 3 | 1 | 1 | 7 | 8 | 8 | 3 | 4 | 10 | 46
    2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-Emergent Adverse Event (TEAE) and as Per the Severity
Description: AE is defined as any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. A treatment-emergent AE is any AE either reported for first time or worsening of a pre-existing event after the first dose of study drug. Grade 1 AEs is defined as Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 AEs is defined as Moderate; minimal, local, or non-invasive intervention indicated; limiting age-appropriate activities of daily living. Grade 3 AEs is defined as the severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living and Grade 4 AEs as life-threatening consequences; urgent intervention indicated. Data is reported for Grade 3 and higher severity for this outcome measure.
Time Frame: From screening through 60 days after end of treatment, up to Month 15
Population: The full analysis set (FAS) included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: 0.03 mg/kg Q2W: Participants received IV infusion of study drug at a dose of 0.03 mg/kg Q2W starting on Day 1 of each cycle for up to 15 months.
Arm/Group | Phase 1: 0.03 mg/kg Q2W | Phase 1: 0.1 mg/kg Q2W | Phase 1: 0.3 mg/kg Q2W | Phase 1: 1.0 mg/kg Q2W | Phase 1: 3.0 mg/kg Q2W | Phase 1: 5.0 mg/kg Q2W | Phase 1: 10.0 mg/kg Q2W | Phase 1: 20.0 mg/kg Q2W | Phase 1: 400 mg Q4W | Phase 2: 300 mg Q2W
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 15 | 18 | 16 | 4 | 10 | 22
Participants
  TEAEs | 4 | 4 | 4 | 3 | 15 | 18 | 16 | 4 | 10 | 22
  Grade 3 and Higher | 3 | 3 | 1 | 2 | 8 | 11 | 9 | 3 | 3 | 14

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Day 1 of Cycles 1 and 6 post-dose
Population: The pharmacokinetic (PK) evaluable population included all participants who received at least 1 dose of study drug and provided at least 1 post dose sample (1 PK measurement).
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/mL)
Arm/Group | Phase 1: 0.03 mg/kg Q2W | Phase 1: 0.1 mg/kg Q2W | Phase 1: 0.3 mg/kg Q2W | Phase 1: 1.0 mg/kg Q2W | Phase 1: 3.0 mg/kg Q2W | Phase 1: 5.0 mg/kg Q2W | Phase 1: 10.0 mg/kg Q2W | Phase 1: 20.0 mg/kg Q2W | Phase 1: 400 mg Q4W | Phase 2: 300 mg Q2W
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 15 | 18 | 16 | 4 | 10 | 22
nanograms per millilitre (ng/mL)
  Cycle 1 (After the First Dose): number analyzed (Participants) | 4 | 4 | 4 | 3 | 15 | 15 | 14 | 4 | 8 | 21
  Cycle 1 (After the First Dose) | 781 (135) | 2700 (779) | 6450 (1330) | 21,600 (321) | 66,000 (13,700) | 128,000 (30,100) | 283,000 (71,500) | 437,000 (60,500) | 127,000 (25,400) | 103,000 (25,600)
  Cycle 6: number analyzed (Participants) | 0 | 0 | 2 | 1 | 5 | 5 | 3 | 0 | 3 | 7
  Cycle 6 |  |  | 7420 (573) | 36,500 (NA) — Standard deviation was not estimable due to low number of participants analyzed. | 107,000 (25,500) | 176,000 (65,700) | 409,000 (97,000) |  | 168,000 (28,500) | 137,000 (21,900)

3. Secondary Outcome: Time to Maximum Concentration (Tmax)
Time Frame: Day 1 of Cycles 1 and 6 post-dose
Population: The PK evaluable population included all participants who received at least 1 dose of study drug and provided at least 1 post dose sample (1 PK measurement).
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Phase 1: 0.03 mg/kg Q2W | Phase 1: 0.1 mg/kg Q2W | Phase 1: 0.3 mg/kg Q2W | Phase 1: 1.0 mg/kg Q2W | Phase 1: 3.0 mg/kg Q2W | Phase 1: 5.0 mg/kg Q2W | Phase 1: 10.0 mg/kg Q2W | Phase 1: 20.0 mg/kg Q2W | Phase 1: 400 mg Q4W | Phase 2: 300 mg Q2W
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 15 | 18 | 16 | 4 | 10 | 22
hours (hr)
  Cycle 1 (After the First Dose): number analyzed (Participants) | 4 | 4 | 4 | 3 | 15 | 15 | 14 | 4 | 8 | 21
  Cycle 1 (After the First Dose) | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 4.0] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 4.0] | 0.1 [0.1 to 4.0] | 0.1 [0.1 to 4.0] | 0.1 [0.1 to 4.0] | 0.1 [0.1 to 4.0] | 0.1 [0.1 to 4.0]
  Cycle 6: number analyzed (Participants) | 0 | 0 | 2 | 1 | 5 | 5 | 3 | 0 | 3 | 7
  Cycle 6 |  |  | 0.1 [0.1 to 0.1] | 4.0 [NA to NA] — Lower and upper limits were not estimable due to low number of participants analyzed. | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 4.0] | 0.1 [0.1 to 4.0] |  | 0.1 [0.1 to 4.0] | 0.1 [0.1 to 4.0]

4. Secondary Outcome: Minimum Observed Plasma Concentration Over the Dose Interval (Cmin)
Time Frame: Day 1 of Cycles 2, 3, 4, 6, and 7 post-dose
Population: The PK evaluable population included all participants who received at least 1 dose of study drug and provided at least 1 post dose sample (1 PK measurement). Data is presented for those cycles for which data is available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1: 0.03 mg/kg Q2W | Phase 1: 0.1 mg/kg Q2W | Phase 1: 0.3 mg/kg Q2W | Phase 1: 1.0 mg/kg Q2W | Phase 1: 3.0 mg/kg Q2W | Phase 1: 5.0 mg/kg Q2W | Phase 1: 10.0 mg/kg Q2W | Phase 1: 20.0 mg/kg Q2W | Phase 1: 400 mg Q4W | Phase 2: 300 mg Q2W
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 15 | 18 | 16 | 4 | 10 | 22
ng/mL
  Cycle 2: number analyzed (Participants) | 4 | 3 | 4 | 3 | 12 | 17 | 16 | 4 | 8 | 19
  Cycle 2 | 42.1 (48.8) | 460 (131) | 1110 (762) | 4910 (1420) | 14,800 (6160) | 25,600 (12,100) | 58,000 (23,900) | 95,400 (33,300) | 13,000 (10,100) | 22,800 (5880)
  Cycle 3: number analyzed (Participants) | 2 | 3 | 4 | 2 | 11 | 17 | 13 | 3 | 6 | 18
  Cycle 3 | 0.0 (0.0) | 206 (187) | 900 (1050) | 8290 (5530) | 23,500 (10,600) | 36,200 (25,500) | 89,200 (35,000) | 117,000 (44,400) | 22,800 (10,200) | 36,800 (16,300)
  Cycle 4: number analyzed (Participants) | 2 | 3 | 4 | 1 | 10 | 12 | 10 | 2 | 5 | 13
  Cycle 4 | 0.0 (0.0) | 29.1 (50.5) | 1390 (1230) | 10,300 (NA) — Standard deviation could not be calculated for single patient | 25,700 (15,000) | 46,700 (36,500) | 135,000 (73,700) | 135,000 (66,300) | 20,500 (11,200) | 31,600 (15,200)
  Cycle 6: number analyzed (Participants) | 1 | 1 | 4 | 1 | 7 | 6 | 6 | 0 | 3 | 10
  Cycle 6 | 0.0 (0.0) | 0.0 (0.0) | 1210 (1260) | 15,100 (NA) — Standard deviation could not be calculated for single patient | 34,900 (19,000) | 71,800 (42,800) | 133,000 (33,200) |  | 21,300 (14,100) | 42,400 (15,600)
  Cycle 7: number analyzed (Participants) | 0 | 1 | 4 | 1 | 5 | 6 | 5 | 0 | 3 | 7
  Cycle 7 |  | 0.0 (0.0) | 939 (1060) | 15,500 (NA) — Standard deviation could not be calculated for single patient | 41,100 (16,700) | 64,900 (34,800) | 124,000 (42,100) |  | 27,500 (18,300) | 63,400 (53,500)

5. Secondary Outcome: Area Under the Plasma Time Curve From Time = 0 to the Last Measurable Concentration (AUC0-t)
Time Frame: Day 1 of Cycles 1 and 6 post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microgram (μg)*hr/mL
Arm/Group | Phase 1: 0.03 mg/kg Q2W | Phase 1: 0.1 mg/kg Q2W | Phase 1: 0.3 mg/kg Q2W | Phase 1: 1.0 mg/kg Q2W | Phase 1: 3.0 mg/kg Q2W | Phase 1: 5.0 mg/kg Q2W | Phase 1: 10.0 mg/kg Q2W | Phase 1: 20.0 mg/kg Q2W | Phase 1: 400 mg Q4W | Phase 2: 300 mg Q2W
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 15 | 18 | 16 | 4 | 10 | 22
microgram (μg)*hr/mL
  Cycle 1 (After the First Dose): number analyzed (Participants) | 4 | 4 | 4 | 3 | 15 | 15 | 14 | 4 | 8 | 21
  Cycle 1 (After the First Dose) | 70.7 (29.0) | 302 (115) | 850 (108) | 3130 (254) | 8880 (2710) | 17,900 (4970) | 39,800 (10,300) | 67,500 (7920) | 25,400 (10,000) | 13,400 (3520)
  Cycle 6: number analyzed (Participants) | 0 | 0 | 2 | 1 | 5 | 5 | 3 | 0 | 3 | 7
  Cycle 6 |  |  | 1070 (392) | 7190 (NA) — Standard deviation was not estimable due to low number of participants analyzed. | 16,200 (10,000) | 33,700 (17,400) | 79,000 (13,400) |  | 42,100 (19,500) | 22,000 (6640)

6. Secondary Outcome: Objective Response Rate (ORR) Per RECIST v1.1 and Modified RECISTv1.1 (mRECIST)
Description: ORR is defined as the percentage of participants having complete response (CR) or partial response (PR), as determined by investigator assessment of radiographic disease assessments. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
Time Frame: Baseline and every 8 weeks for the first 12 months and then every 12 weeks thereafter up to 15 months
Population: The FAS included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: 0.03 mg/kg Q2W | Phase 1: 0.1 mg/kg Q2W | Phase 1: 0.3 mg/kg Q2W | Phase 1: 1.0 mg/kg Q2W | Phase 1: 3.0 mg/kg Q2W | Phase 1: 5.0 mg/kg Q2W | Phase 1: 10.0 mg/kg Q2W | Phase 1: 20.0 mg/kg Q2W | Phase 1: 400 mg Q4W | Phase 2: 300 mg Q2W
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 15 | 18 | 16 | 4 | 10 | 22
percentage of participants
  RECIST v1.1 | 0.0 | 0.0 | 25.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 4.5
  mRECIST v1.1 | 0.0 | 0.0 | 25.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

7. Secondary Outcome: Duration of Response (DOR) Per RECIST and mRECIST
Description: DOR is defined as the time from earliest date of disease response (CR or PR) until earliest date of disease progression, as determined by investigator assessment of radiographic disease assessments per RECIST v1.1 and mRECIST, or death due to any cause if occurring sooner than progression. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
Time Frame: Baseline and every 8 weeks for the first 12 months and then every 12 weeks thereafter up to 15 months
Population: The FAS included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 1: 0.03 mg/kg Q2W | Phase 1: 0.1 mg/kg Q2W | Phase 1: 0.3 mg/kg Q2W | Phase 1: 1.0 mg/kg Q2W | Phase 1: 3.0 mg/kg Q2W | Phase 1: 5.0 mg/kg Q2W | Phase 1: 10.0 mg/kg Q2W | Phase 1: 20.0 mg/kg Q2W | Phase 1: 400 mg Q4W | Phase 2: 300 mg Q2W
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 15 | 18 | 16 | 4 | 10 | 22
Days
  RECIST v1.1 | NA [NA to NA] — There were no participants with response at given timepoint thus median and 95% CI was not estimable. | NA [NA to NA] — There were no participants with response at given timepoint thus median and 95% CI was not estimable. | 169.0 [NA to NA] — Lower and upper limits of 95% CI were not estimable as there were not enough participants with response | NA [NA to NA] — There were no participants with response at given timepoint thus median and 95% CI was not estimable. | NA [NA to NA] — There were no participants with response at given timepoint thus median and 95% CI was not estimable. | NA [NA to NA] — There were no participants with response at given timepoint thus median and 95% CI was not estimable. | NA [NA to NA] — There were no participants with response at given timepoint thus median and 95% CI was not estimable. | NA [NA to NA] — There were no participants with response at given timepoint thus median and 95% CI was not estimable | NA [NA to NA] — There were no participants with response at given timepoint thus median and 95% CI was not estimable | NA [NA to NA] — There was 1 participant with response, but DOR was ongoing at time of censoring, which was 399 days after initial response.
  mRECIST v1.1 | NA [NA to NA] — There were no participants with response at given timepoint thus median and 95% CI was not estimable. | NA [NA to NA] — There were no participants with response at given timepoint thus median and 95% CI was not estimable. | 169.0 [NA to NA] — Lower and upper limits of 95% CI were not estimable as there were not enough participants with response | NA [NA to NA] — There were no participants with response at given timepoint thus median and 95% CI was not estimable. | NA [NA to NA] — There were no participants with response at given timepoint thus median and 95% CI was not estimable. | NA [NA to NA] — There were no participants with response at given timepoint thus median and 95% CI was not estimable. | NA [NA to NA] — There were no participants with response at given timepoint thus median and 95% CI was not estimable. | NA [NA to NA] — There were no participants with response at given timepoint thus median and 95% CI was not estimable. | NA [NA to NA] — There were no participants with response at given timepoint thus median and 95% CI was not estimable. | NA [NA to NA] — There was 1 participant with response, but DOR was ongoing at time of censoring, which was 399 days after initial response.

8. Secondary Outcome: Duration of Disease Control Per RECIST and mRECIST
Description: Duration of disease control (CR, PR, and stable disease [SD]), as measured from first report of SD or better until disease progression, as determined by investigator assessment of radiographic disease assessments per RECIST v1.1 and mRECIST, or death due to any cause if occurring sooner than progression. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Baseline and every 8 weeks for the first 12 months and then every 12 weeks thereafter up to 15 months
Population: The FAS included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1: 0.03 mg/kg Q2W | Phase 1: 0.1 mg/kg Q2W | Phase 1: 0.3 mg/kg Q2W | Phase 1: 1.0 mg/kg Q2W | Phase 1: 3.0 mg/kg Q2W | Phase 1: 5.0 mg/kg Q2W | Phase 1: 10.0 mg/kg Q2W | Phase 1: 20.0 mg/kg Q2W | Phase 1: 400 mg Q4W | Phase 2: 300 mg Q2W
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 15 | 18 | 16 | 4 | 10 | 22
days
  RECIST v1.1 | NA [NA to NA] — There were no participants with stable disease or response at given timepoint thus median and 95% CI was not estimable. | NA [NA to NA] — There were no participants with stable disease or response at given timepoint thus median and 95% CI was not estimable | 169.0 [NA to NA] — Lower and upper limits of 95% CI were not estimable as there were not enough participants with stable disease or response | 91.0 [NA to NA] — Lower and upper limits of 95% CI were not estimable as there were not enough participants with stable disease or response | 58.5 [36.0 to 226.0] | 58.0 [53.0 to 109.0] | 62.0 [59.0 to 113.0] | 61.0 [NA to NA] — Lower and upper limits of 95% CI were not estimable as there were not enough participants with stable disease or response | 113.0 [15.0 to 172.0] | 213.0 [54.0 to NA] — Upper limit of 95% CI was not estimable as there were not enough participants with stable disease or response.
  mRECIST v1.1 | NA [NA to NA] — There were no participants with stable disease or response at given timepoint thus median and 95% CI was not estimable | NA [NA to NA] — There were no participants with stable disease or response at given timepoint thus median and 95% CI was not estimable | 169.0 [NA to NA] — Lower and upper limits of 95% CI were not estimable as there were not enough participants with stable disease or response | 91.0 [NA to NA] — Lower and upper limits of 95% CI were not estimable as there were not enough participants with stable disease or response | 58.5 [36.0 to 226.0] | 58.0 [53.0 to 109.0] | 62.0 [59.0 to 113.0] | 61.0 [NA to NA] — Lower and upper limits of 95% CI were not estimable as there were not enough participants with stable disease or response | 113.0 [15.0 to 172.0] | 213.0 [54.0 to NA] — Upper limit of 95% CI was not estimable as there were not enough participants with stable disease or response.

9. Secondary Outcome: Progression Free Survival (PFS) Per RECIST and mRECIST
Description: PFS is defined as the time from date of first dose of study drug until the earliest date of disease progression, as determined by investigator assessment of objective radiographic disease assessments per RECIST v1.1 and mRECIST, or death due to any cause if occurring sooner than progression. Progression is defined by RECIST and mRECIST as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study and an absolute lesion increase of at least 5 mm or the appearance of new lesions.
Time Frame: Baseline and every 8 weeks for the first 12 months and then every 12 weeks thereafter up to 15 months
Population: The FAS included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: 0.03 mg/kg Q2W | Phase 1: 0.1 mg/kg Q2W | Phase 1: 0.3 mg/kg Q2W | Phase 1: 1.0 mg/kg Q2W | Phase 1: 3.0 mg/kg Q2W | Phase 1: 5.0 mg/kg Q2W | Phase 1: 10.0 mg/kg Q2W | Phase 1: 20.0 mg/kg Q2W | Phase 1: 400 mg Q4W | Phase 2: 300 mg Q2W
Number analyzed (Participants) | 4 | 4 | 4 | 3 | 15 | 18 | 16 | 4 | 10 | 22
months
  PFS under RECIST v1.1 | 1.64 [0.89 to 1.84] | 1.84 [0.53 to 1.84] | 6.70 [1.64 to 11.04] | 1.48 [1.18 to 4.70] | 1.87 [0.72 to 3.68] | 1.87 [1.48 to 3.61] | 1.84 [0.95 to 3.58] | 2.78 [0.76 to 3.75] | 2.14 [1.74 to 5.55] | 1.87 [1.68 to 3.61]
  PFS under mRECIST v1.1 | 1.64 [0.89 to 1.84] | 1.84 [0.53 to 1.84] | 6.70 [1.64 to 11.04] | 1.48 [1.18 to 4.70] | 1.87 [0.72 to 3.68] | 1.87 [1.48 to 3.61] | 1.84 [0.95 to 3.58] | 2.78 [0.76 to 3.75] | 2.14 [1.74 to 5.55] | 1.87 [1.68 to 3.61]

ADVERSE EVENTS:
Time Frame: From screening through 60 days after end of treatment, up to Month 15
Groups:
- Total: Total
Arm/Group | Phase 1: 0.03 mg/kg Q2W | Phase 1: 0.1 mg/kg Q2W | Phase 1: 0.3 mg/kg Q2W | Phase 1: 1.0 mg/kg Q2W | Phase 1: 3.0 mg/kg Q2W | Phase 1: 5.0 mg/kg Q2W | Phase 1: 10.0 mg/kg Q2W | Phase 1: 20.0 mg/kg Q2W | Phase 1: 400 mg Q4W | Phase 2: 300 mg Q2W | Total
All-Cause Mortality (participants affected / at risk) | 2/4 | 3/4 | 1/4 | 1/3 | 4/15 | 5/18 | 3/16 | 1/4 | 1/10 | 5/22 | 26/100
Serious Adverse Events (participants affected / at risk) | 3/4 | 3/4 | 1/4 | 2/3 | 6/15 | 6/18 | 7/16 | 2/4 | 3/10 | 10/22 | 43/100
Other Adverse Events (participants affected / at risk) | 4/4 | 3/4 | 4/4 | 3/3 | 15/15 | 18/18 | 16/16 | 4/4 | 10/10 | 22/22 | 99/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: 0.03 mg/kg Q2W (N=4) | Phase 1: 0.1 mg/kg Q2W (N=4) | Phase 1: 0.3 mg/kg Q2W (N=4) | Phase 1: 1.0 mg/kg Q2W (N=3) | Phase 1: 3.0 mg/kg Q2W (N=15) | Phase 1: 5.0 mg/kg Q2W (N=18) | Phase 1: 10.0 mg/kg Q2W (N=16) | Phase 1: 20.0 mg/kg Q2W (N=4) | Phase 1: 400 mg Q4W (N=10) | Phase 2: 300 mg Q2W (N=22) | Total (N=100)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 5 (5)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 10 (10)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perforation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombotic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: 0.03 mg/kg Q2W (N=4) | Phase 1: 0.1 mg/kg Q2W (N=4) | Phase 1: 0.3 mg/kg Q2W (N=4) | Phase 1: 1.0 mg/kg Q2W (N=3) | Phase 1: 3.0 mg/kg Q2W (N=15) | Phase 1: 5.0 mg/kg Q2W (N=18) | Phase 1: 10.0 mg/kg Q2W (N=16) | Phase 1: 20.0 mg/kg Q2W (N=4) | Phase 1: 400 mg Q4W (N=10) | Phase 2: 300 mg Q2W (N=22) | Total (N=100)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 3 (4) | 8 (9) | 2 (2) | 2 (2) | 1 (1) | 22 (25)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Affect lability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 8 (8)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 1 (2) | 4 (4) | 15 (16)
Anhedonia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 8 (8)
Asthenia (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 9 (10)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 10 (10)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breath odour (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Clubbing (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 13 (15)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 3 (3) | 2 (3) | 3 (3) | 4 (4) | 20 (21)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 9 (10)
Denture wearer (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 3 (4) | 4 (7) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 15 (20)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 6 (6)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (7) | 4 (4) | 3 (3) | 1 (1) | 3 (4) | 5 (5) | 24 (26)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 5 (5) | 7 (8) | 2 (2) | 5 (5) | 11 (12) | 38 (40)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 7 (7)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Globulins increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Grip strength decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 12 (13)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 8 (8)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 3 (5)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (3) | 7 (8)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 7 (7)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Local swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 5 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 7 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 3 (3) | 5 (6) | 6 (7) | 1 (1) | 2 (2) | 5 (6) | 24 (29)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 5 (6) | 0 (0) | 1 (1) | 1 (1) | 5 (6) | 16 (18)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (5)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericarditis constrictive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 6 (6)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural discharge (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 5 (6) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 17 (19)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 8 (8)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 2 (4) | 5 (5) | 0 (0) | 1 (1) | 4 (4) | 19 (22)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 8 (12)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 6 (7)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Systemic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 6 (7)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 5 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 3 (5) | 3 (3) | 5 (5) | 2 (3) | 1 (1) | 2 (2) | 19 (24)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT02697591/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT02697591/SAP_001.pdf